CLINICAL TRIAL: NCT02680119
Title: An Open Label, Randomized, 2-Period, 2-Treatment,2-Sequence, Crossover, Single-Dose BE Study of Esomeprazole Mg DR Capsule 40 mg [Torrent] Versus Nexium [AastraZeneca]- Sprinkled Over Apple Sauce in Subjects-Fasting Condition
Brief Title: BE of Torrent's Esomeprazole Mg DR Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK-10-181
Record Dates: First submitted 2016-02-02; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Torrent's Esomeprazole Magnesium DR Capsules 40 mg
  Interventions: Drug: Torrent's Esomeprazole Magnesium DR Capsules 40 mg
- Reference (Active Comparator): Nexium 40 mg DR Capsules of AstraZeneca LP, USA
  Interventions: Drug: Nexium 40 mg DR Capsules of AstraZeneca LP, USA.

INTERVENTIONS:
Drug: Nexium 40 mg DR Capsules of AstraZeneca LP, USA. — oral, crossover
  Other Names: esomeprazole magnesium delayed release capsules
  Arms: Reference
Drug: Torrent's Esomeprazole Magnesium DR Capsules 40 mg — oral, crossover
  Other Names: esomeprazole magnesium delayed release capsules
  Arms: Test

SUMMARY:
Subjects to compare the single dose bioavailability of Torrent's Esomeprazole Mg DR Capsule 1×40 mg and Nexium 40 mg DR Capsule containing Esomeprazole 40 mg of AastraZeneca LP, USA. Dosing periods of studies were separated by a washout period of 5 days.

DETAILED DESCRIPTION:
An open Label, Randomized, 2-Period, 2-Treatment,2-Sequence, Crossover, Single-Dose Bioequivalence Study of Esomeprazole Mg DR Capsule containing Esomeprazole Mg 40 mg [ Test Formulation, Torrent Pharmaceutical Ltd., India] Versus Nexium 40 mg DR Capsule containing Esomeprazole 40 mg [Reference Formulation, AastraZeneca LP, USA] Under administered as the contents of capsule sprinkled over apple sauce in Healthy Human Volunteers Under Fasting Condition.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* Age: 18-45 years
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day.

Exclusion Criteria:

* Inability to communicate or co-operate.
* Administration of any study drug in the period 0 to 3 months before entry to the study,
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of pre-existing bleeding disorder.
* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* HIV, HCV, HBsAg positive volunteers.
* History of alcohol or drug abuse.
* History of consumption of prescribed medication since last 14days or OTC medication/ herbal remedies since last 7 days before beginning of the study.
* Positive to Breath alcohol test.
* Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, Cocaine positive volunteers based on urine test.
* Systolic blood pressure less than 100 mmHg or more than 140 mmHg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°F or more than 98.6°F.
* Respiratory rate less than 12/minute or more than 20/minute.
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* Recent History of kidney or liver dysfunction.
* Volunteers suffering from any psychiatric (acute or chronic) disorder.
* Existence of any surgical or medical condition, which, in the judgment of the Chief Investigator and/or clinical investigator/physician, might interfere with the absorption; distribution,· metabolism or excretion of the drug or likely to compromise the safety of Volunteers.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose to 20 hour post dose
  Pharmacokinetic Evaluation
AUC | Pre-dose to 20 hour post dose
  Pharmacokinetic Evaluation

IPD SHARING:
Plan to Share IPD: No